CLINICAL TRIAL: NCT02704780
Title: Umbilical Vein Injection of 800µg Misoprostol Versus 400 µg Misoprostol in the Treatment of Retained Placenta: A Multicenter, Randomized Double Blind Controlled Trial
Brief Title: Two Different Regimens of Misoprostol in Retained Placenta
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Shahla Alalaf, Professor Shahla K.Alalaf, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HawlerMU
Record Dates: First submitted 2016-02-19; First posted 2016-03-10 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Postpartum Haemorrhage; Retained Placenta
Keywords: Retained placenta; Misoprostol; double blind; Randomization; Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage; Placenta, Retained; Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 400 Microgram Misoprostol (Active Comparator): Misoprostol 400 micro-gram dissolved in 20 mL normal saline will be injected in the umbilical vein in the first group
  Interventions: Drug: Misoprostol
- 800 Microgram Misoprostol (Active Comparator): Misoprostol 800 micro-gram dissolved in 20 mL normal saline will be injected in umbilical cord of the second group
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 2 regimes of misoprostol 400 microgram and 800 microgram injections used for 2 groups of women
  Other Names: Cytotic

SUMMARY:
This study evaluates intra umbilical vein injection of 800 µg versus 400 µg misoprostol for the treatment of retained placenta to reduce the need of manual removal of placenta under general anaesthesia

DETAILED DESCRIPTION:
The third stage of labor may be complicated by retained placenta, which may cause severe bleeding and infection, with a potentially fatal outcome. Manual removal of placenta is the current standard of management of retained placenta which usually requires general or regional anaesthesia at a hospital and it is an invasive procedure that may lead to bleeding, trauma and infection. Intraumbilical injection of uterotonic agent( misoprostol) is an easy, non invasive procedure. A randomized clinical trial are required to determine the difference between two doses of misoprostol 400 versus 800 micro gram for management of retained placenta

ELIGIBILITY:
Inclusion Criteria:

* women with a singleton pregnancy, delivered vaginally
* 28 weeks of gestation and more,
* had a prolonged third stage of labor (more than 30 minutes) despite active management,
* Haemodynamically stable and accept to participate in the trial

Exclusion Criteria:

* multiple pregnancies,
* previous caesarean delivery,
* haemodynamically instability, severe anaemia (haemoglobin concentration <8 g/dL),
* chorioamnionitis
* Refused to participate in the trial

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 509 (Actual)
Dates: Start 2016-03; Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Delivery of placenta after injection of of 400 Microgram intraumbilical misoprostol versus 800 microgram of misoprostol | up to 30 minutes after intraumbilical injection
  complete delivery of placenta after injection of intraumbilical misoprostol

SECONDARY OUTCOMES:
The amount of blood loss vaginally in both groups | up to 30 minutes after injection of placenta
  To estimate the amount of vaginal blood loss from time of injection of the the interventional drug and till the delivery of the placenta
The time of delivery of placenta in both groups | up to 30 minutes after delivery of the placenta
  the time interval estimation from the injection to complete delivery of the placenta
side effects of misoprostol | up to 24 hours after delivery of placenta
  Any side effects related to misoprostol after the injection (Fever, severing , diarrhea)

CONTACTS AND LOCATIONS:
Overall Officials: Shahla K. Alalaf, professor, Principal Investigator — Hawler Medical University; Namir G. Al Tawil, Professor, Study Director — Hawler Medical University; Ariana Kh. Jawad, Assistant professor, Study Chair — KBMS; Bahar Q. Muhammad, CABOG, Study Chair — Maternity Teaching Hospital; Jinan N. Hassan, IBMS, Study Chair — Duhok university; Salim A. Salim, Master, Study Chair — Al-Azhar University; Khalida M. Ameen, CABOG, Study Chair — Karkuk Medical college; Maryam B. Mahmood, FICOG, Study Chair — Sulaimani Maternity Hospital; Khansa H. Abdul Rahman, MBChB, Study Chair — Maternity Teaching Hospital
Locations (1):
- Hawler Medical university, Erbil, Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumar N, Jahanfar S, Haas DM, Weeks AD. Umbilical vein injection for management of retained placenta. Cochrane Database Syst Rev. 2021 Mar 11;3(3):CD001337. doi: 10.1002/14651858.CD001337.pub3. PMID 33705565